CLINICAL TRIAL: NCT05781308
Title: A Non-comparative Randomized Phase II Trial Evaluating the Combination of Paclitaxel-bevacizumab ± Atezolizumab in Patients With Advanced Non-squamous NSCLC Progressing After Immunotherapy and Chemotherapy
Brief Title: Combination of Paclitaxel-bevacizumab ± Atezolizumab in Patients With Advanced NSCLC Progressing After Immunotherapy & Chemotherapy
Acronym: ADAPTABLE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-2201
Record Dates: First submitted 2023-02-17; First posted 2023-03-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: IFCT; NCSLC; atezolizumab; immunotherapy; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Bevacizumab; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: paclitaxel + bevacizumab (Other): Bevacizumab 15 mg/kg and paclitaxel 200 mg/m² intravenously every three weeks until progression.
  Interventions: Drug: Paclitaxel; Drug: Bevacizumab
- Arm B: paclitaxel + bevacizumab + atezolizumab (Experimental): Atezolizumab 1200 mg, bevacizumab 15 mg/kg and paclitaxel 200 mg/m² intravenously every three weeks until progression.
  Interventions: Drug: Paclitaxel; Drug: Bevacizumab; Drug: Atezolizumab

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 200 mg/m² every 3 weeks
Drug: Bevacizumab — Bevacizumab 15 mg/kg every 3 weeks
  Other Names: Avastin
Drug: Atezolizumab — 1200 mg every 3 weeks
  Other Names: Tecentriq
  Arms: Arm B: paclitaxel + bevacizumab + atezolizumab

SUMMARY:
This is an open-label, randomized, non-comparative, multicentre, phase II study in which NSCLC patients who have progressed following chemotherapy and immunoptherapy are randomized to receive treatment with either paclitaxel and bevacizumab (Arm A), or paclitaxel, bevacizumab and atezolizumab (Arm B). An estimated 156 patients (52 in Arm A, 104 in Arm B) will be enrolled at approximately 40 centres. Patients will be treated until disease progression, unacceptable toxicity, withdrawal of consent or another discontinuation criterion is met. For patients in Arm B, continuation of atezolizumab beyond progression is permitted, at the investigator's discretion, if there is evidence of continued clinical benefit. The null hypothesis is progression free survival at 6 months ≤ 50% for Arm B, which is considered not sufficiently clinically meaningful to warrant further study. The alternative hypothesis is that 66% or more of patients in Arm B would achieve progression free survival at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal patient care.

   Patients must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing.
2. Male or female aged at least 18 years old.
3. ECOG Performance Status of 0 or 1.
4. Histologically or cytologically documented locally advanced unresectable NSCLC (i.e. stage IIIB/IIIC not eligible for definitive chemo-radiotherapy) or metastatic NSCLC (i.e. Stage IV) (per the 8th edition of Union Internationale Contre le Cancer/American Joint Committee on Cancer [UICC/AJCC] staging system) of non-squamous histology.

   Note: patients with tumours of mixed histology must be classified as non-squamous or squamous based on the major histological component.
5. Patients progressing after treatment with immunotherapy (anti-PD-1 or anti-PD-L1 Ab) and a doublet of platinum-based chemotherapy, given concomitantly or sequentially to the exclusion of any other treatment.
6. Patients without contraindications to bevacizumab.
7. The investigator must confirm prior to enrolment that the patient has adequate tumour tissue available. Tumour biopsy should be exploitable for molecular analysis.

   Note: Tumour tissue collected after the patient was diagnosed with metastatic disease is preferred.

   Tumour tissue sample must not be from previously radiated locations. Tumour sample must be one block or at least 10 unstained slides of analysable tissue.

   If archival tissue is either insufficient or unavailable, the patient may still be eligible upon discussion with IFCT.
8. All patients must have at least one measurable target lesion according to RECIST v1.1. Previously irradiated lesions can only be considered measurable disease if disease progression has been unequivocally documented at that site since radiation and the previously irradiated lesion is not the only site of measurable disease.
9. Life expectancy ≥ 12 weeks
10. Adequate hematologic and end-organ function, defined by the following laboratory test results:

    * ANC ≥ 1500 cells/µL (without granulocyte colony-stimulating factor support within 14 days prior to C1D1).
    * WBC count ≥ 2500/µL.
    * Lymphocyte count ≥ 500/µL.
    * Platelet count ≥ 100 000/µL (without transfusion within 14 days prior to C1D1).
    * Haemoglobin ≥ 9.0 g/dL (patients may be transfused or receive erythropoietic treatment as per local standard of care).
    * Total bilirubin ≤ 1.5 x upper limit of normal (ULN).
    * Patients with known Gilbert's disease or hepatic metastasis who have serum bilirubin level ≤ 3 x ULN may be enrolled.
    * AST and ALT ≤ 3 x ULN, with the following exception: patients with documented liver metastases: AST and ALT ≤ 5 x ULN; ALP ≤ 2.5 x ULN; or patients with documented bone metastases: ALP ≤ 5 x ULN.
    * Serum albumin ≥ 2.5 g/dL.
    * aPTT or PTT and PT or INR ≤ 1.5 x ULN. This applies only to patients who are not receiving therapeutic anticoagulation. Patients receiving therapeutic anticoagulation should be on a stable dose for at least 1 week prior to C1D1.
11. Measured or calculated creatinine clearance ≥ 50 mL/min calculated using the local standard method.
12. Recovered from all toxicities associated with prior treatment, to acceptable baseline status, or NCI CTCAE v5.0 Grade 0 or 1, except for toxicities not considered a safety risk, such as alopecia or vitiligo. According to national (FITC) and international recommendations, certain severe immuno-induced toxicities are absolute exclusion criteria for the (re)introduction of anti-PD-L1 antibodies (atezolizumab) (e.g. pneumopathy, colitis etc.). If in doubt, please contact the IFCT.
13. For women of childbearing potential (including women who have had a tubal ligation), serum pregnancy test must be performed and documented as negative within 14 days prior to C1D1.
14. Women of childbearing potential must remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 6 months after the last dose of study drugs. Women must refrain from donating eggs during this same period. A woman is considered to be of childbearing potential if she is post-menarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries or uterus). Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. Hormonal contraceptive methods must be supplemented by a barrier method plus spermicide. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g. calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
15. Men with female partners of childbearing potential or pregnant female partners, must remain abstinent or use a condom during the treatment period and for at least 6 months after the last dose of study treatment to avoid exposing the embryo. Men must refrain from donating sperm during this same period. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g. calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
16. Participant has national health insurance coverage.

Exclusion Criteria:

1. Known molecular alteration of EGFR, ALK, ROS1, RET, NTRK, MET, NRG1.
2. Patients previously treated by bevacizumab combined with first-line chemotherapy for NSCLC.
3. Patients with a previous treatment by taxane (docetaxel, paclitaxel). A patient with a previous treatment by peri-operative taxane or in association with radiotherapy is eligible if the treatment has been stopped for more than 6 months.
4. Patients previously treated for unresectable stage III NSCLC are not eligible if they progressed during or within 6 months of stopping consolidation immunotherapy. Patients previously treated by peri-operative immunotherapy for stage I, II or III NSCLC are not eligible.
5. Patients with symptomatic brain metastasis, leptomeningeal disease or other active CNS metastases are not eligible. Note: patients with previously treated or untreated brain metastases may participate, provided they are stable (e.g. without evidence of progression by radiographic imaging for at least 28 days before the first dose of study treatment and neurologic symptoms have returned to baseline). Patients must have no evidence of new or enlarging brain metastases or CNS oedema. Patients must have discontinued use of steroids (with a dose > 10 mg prednisone equivalent daily) at least 7 days before the first dose of study treatment.
6. Spinal cord compression not definitively treated with surgery or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for ≥ 2 weeks prior to screening.
7. Malignancies other than NSCLC within 3 years prior to randomization, with the exception of those with a negligible risk of metastasis or death, or treated with expected curative outcome (such as adequately treated in situ cervical cancer, basal or squamous cell skin cancer, localized prostate cancer, ductal carcinoma in situ, or stage I uterine cancer).
8. Inability to comply with study or follow-up procedures.
9. Pregnant, lactating, or breastfeeding women.
10. Severe infections (including active tuberculosis) within 4 weeks prior to initiation of study treatment, including but not limited to hospitalization for complications of infection, bacteraemia, or severe pneumonia.
11. Received oral or IV antibiotics (including antifungals) within 2 weeks prior to randomization. Patients receiving prophylactic antibiotics (e.g. for prevention of a urinary tract infection or chronic obstructive pulmonary disease exacerbations) are eligible.
12. Major surgical procedure within 4 weeks prior to randomization, or anticipation of need for a major surgical procedure during the course of the study.
13. Inability to understand the local language (French).
14. Any disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, that may affect the interpretation of the results, or that may render the patient at high risk from treatment complications.
15. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
16. Known hypersensitivity or allergy to Chinese hamster ovary cell products or any component of the atezolizumab formulation.
17. Active or history of autoimmune disease with the following exceptions:

    * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study following discussion with IFCT.
    * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen may be eligible for this study following discussion with IFCT.
    * Patients with benign rheumatoid polyarthritis not needing any immunosuppressive systemic treatment.
    * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g. patients with psoriatic arthritis would be excluded) are permitted provided they meet the following conditions:

      * Rash must cover less than 10% of body surface area (BSA).
      * Disease is well controlled at baseline and only requires low potency topical steroids.
      * No acute exacerbations of the underlying condition within the last 12 months requiring treatment with either PUVA (psoralen plus ultraviolet A radiation), methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral steroids.
18. Prior allogeneic bone marrow transplantation or prior solid organ transplantation.
19. History of idiopathic pulmonary fibrosis (including pneumonitis), organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia), drug induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on chest computed tomography (CT) scan at screening. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
20. Patients with a known history of a positive test for HIV or known AIDS who have not received effective antiretroviral therapy (ART) for the last 4 weeks and who have an HIV viral load >200 copies/mL, regardless of CD4+ T-cell count.
21. Patients with known acute viral hepatitis B or C (HBV, HBC) according to serological tests. Patients with serological sequalae of cured viral hepatitis are eligible.
22. Administration of live, attenuated vaccine within 4 weeks prior to initiation of study treatment or anticipation that such a live attenuated vaccine will be required during the study. Influenza vaccination should be given during influenza season only. Patients must not receive live, attenuated influenza vaccine within 4 weeks prior to enrolment or at any time during the study, and for 5 months following the last study treatment.
23. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone > 10 mg/day, cyclophosphamide, azathioprine, methotrexate, thalidomide, and tumour necrosis factor [TNF-α] antagonists) within 2 weeks prior to randomization. Patients who have received acute, low dose, systemic immunosuppressant medications (e.g. a one-time dose of dexamethasone for nausea) may be eligible for this study following discussion with IFCT. The use of inhaled corticosteroids is allowed. The use of mineralocorticoids (e.g. fludrocortisone) for patients with orthostatic hypotension is allowed. Physiologic doses of corticosteroids for adrenal insufficiency may be allowed after discussion with IFCT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival at 6 months determined by independent reviewer | 6 months after randomization
  PFS is defined as the time between the date of randomization and the first date of documented progression, as determined by independent review, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression Free Survival | At progression, after an average of 15 months.
  PFS is defined as the time between the date of randomization and the first date of documented progression, as determined by investigator, or death due to any cause, whichever occurs first.
Objective Response Rate | At progression, after an average of 15 months.
  ORR is defined as the proportion of patients who have achieved a best overall response of complete response (CR) or partial response (PR) as determined by investigator review of radiographic disease assessments per RECIST v1.1.
Overall Survival | About 39 months
  OS is defined as the time from date of inclusion to the date of death due to any cause. If a death has not been observed by the date of the analysis cut-off, OS will be censored at the date of last contact.
Time until definitive health related quality of life score deterioration | From enrollment to score deterioration, after an average of 15 months.
  The time until definitive health related quality of life score deterioration will be analysed using the EORTC Core Quality of Life Questionnaire (QLQ-C30).
Incidence, nature, and severity of adverse events | From time of informed consent through treatment period and up to 30 days post last dose of study treatment (average of 15 months)]
  Graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0).
Overall health status | At progression, after an average of 15 months.
  Overall health status will also be assessed using the EuroQol 5-dimension 5-level (EQ-5D-5L) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud SCHERPEREEL, Pr, Principal Investigator — Institut Coeur Poumon CHU de Lille; Etienne GIROUX-LEPRIEUR, Pr, Principal Investigator — Pulmonology & Thoracic Oncology Department APHP - Hôpital Ambroise Paré
Locations (44):
- France (44):
  - CHU Amiens, Amiens
  - CHU d'Angers, Angers
  - CH Avignon, Avignon
  - CH Côte Basque, Bayonne
  - CHU Besançon - Hôpital J. MINJOZ, Besançon
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hôpital APHP Ambroise Paré, Boulogne
  - CHU Côte de Nacre, Caen
  - CH Cholet, Cholet
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CH Pasteur, Colmar
  - Centre Hospitalier Intercommunal Créteil CHIC, Créteil
  - Centre Georges-François Leclerc, Dijon
  - CHU Dijon, Dijon
  - Chu Grenoble, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - CH Versailles, Le Chesnay
  - CH Le Mans, Le Mans
  - CHU Lille, Lille
  - CHU Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - APHM Hôpital Nord, Marseille
  - Hôpital Européen, Marseille
  - Hôpitaux Privés de Metz Robert Schuman, Metz
  - GHR Mulhouse et Sud Alsace GHRMSA, Mulhouse
  - CHR Orléans, Orléans
  - Hôpital BICHAT, Paris
  - Hôpital TENON, Paris
  - Groupe Hospitalier Paris Saint Joseph GHPSJ, Paris
  - CH Pau, Pau
  - CHU Bordeaux Haut-Lévèque, Pessac
  - Hospices Civils de Lyon - URCOT, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - CH Annecy Genevois, Pringy
  - CHU Rouen, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - Institut de Cancerologie de l'Ouest ICO, Saint-Herblain
  - Nouvel Hôpital Civil - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - HIA Sainte-Anne, Toulon
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours
  - Clinique Teissier, Valenciennes
  - CH Villefranche Nord Ouest, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data underlying the results reported in this article, as well as the study protocol and statistical analysis plan, will be made available after deidentification immediately following publication and for three years. Researchers who provide a methodologically sound proposal for any purpose may direct proposals to contact@ifct.fr. To gain access, data requestors will need to sign a data access agreement that requires approval by the French Cooperative Thoracic Intergroup.

REFERENCES:
- See also: IFCT website — https://www.ifct.fr/